CLINICAL TRIAL: NCT04925336
Title: Study of Cortical Cerebral Response and Neurovegetative Response to a Nociceptive Stimulus Among Healthy Volunteers
Brief Title: Cerebral and Autonomic Responses to Pain in Healthy Humans
Acronym: ALGOBLOC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL19_0669
Record Dates: First submitted 2020-01-22; First posted 2021-06-14 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Nociceptive Pain; Anesthesia; Healthy
Keywords: Nociceptive stimulation; Healthy volunteer; Simultaneous cortical activation; Neuro-vegetative response
MeSH Terms: conditions — Nociceptive Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Nociceptive intervention arm
  Interventions: Other: Nociceptive stimulation

INTERVENTIONS:
Other: Nociceptive stimulation — These investigations in healthy volunteers will study the association between cerebral and neurovegetative (sympathetic and parasympathetic) electrophysiological responses in response to a controlled and tolerable pain stimulus, determined for each individual. The pain stimulus will be delivered using an electrically conductive glove used in clinical practice for transcutaneous therapeutic stimulation.
  The thresholds of nociception and tolerance will be determined in each healthy volunteer.

SUMMARY:
Evaluating the intraoperative pain is a major challenge for the anesthesia team. During anesthesia, changes in heart rate and blood pressure are interpreted qualitatively to evaluate the sympathetic response to nociceptive stimulation or the adaptation of analgesia during surgery. The new nociception monitors under development quantitatively explore other variables dependent on sympathetic activity or sympathetic / parasympathetic balance, such as the pulse wave amplitude measurement (Surgical Pleth Index (SPI index)), the pupil dilation reflex, respiratory sinus arrhythmia (ANI, Analgesia Nociception Index), or skin conductance index. Taken independently, these tools provide an assessment of nociception based on variations in the autonomic system, more robust than simply observing heart rate or blood pressure raw values.

However, the relationship between variations in the neurovegetative system and pain can be compromised by various factors or intraoperative events such as hypovolemia, bleeding, certain sympathomimetic or sympatholytic treatments, the hypnosis depth, ventilation variation, fast filling, or body temperature. Moreover, investigators do not know the delay between the application of the painful stimulus and the observation of the variation of the different neurovegetative variables. This constitutes a limit of the practitioners' confidence in these monitoring tools.

The nociception transmission pathways of to the vegetative centers and cortical areas are complex. Investigators hypothesis is that neurovegetative variations in response to nociceptive stimulation are not always associated with a cortical somatosensory response. In this project investigators investigate the relation between cortical (EEG) and vegetative reactions to acute and tonic nociceptive stimuli, as a preliminary step to apply these procedures to assess intraoperative reactions to nociceptive procedures in anesthetized patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer over 18 years old
* signed informed consent
* affiliated to a social security

Exclusion Criteria:

* Chronic pathology requiring chronic treatment
* Cardiac rhythm disorders, pacemaker, cardiotropic treatment
* Taking opioid analgesics during the previous week
* Painful chronic, or migraine
* Pathology of the hand, acrosyndrome, carpal tunnel syndrome
* Pregnancy
* People placed under protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Simultaneous scheme of cortical activation and neuro-vegetative responses to controlled nociceptive stimuli | Day 1
  Simultaneous scheme of cortical activation and neuro-vegetative responses secondary to controlled nociceptive stimuli will be defined as the occurrence of at least one among the following:
  * Changes of time-frequency distribution of the electroencephalographic activity during phasic or tonic pain stimulation, compared to a prior baseline period.
  * Recording of cortical evoked responses during phasic pain stimulation in a time latency range between 100-500 msec.
  * Changes in parasympathetic tone measured by Analgesia/Nociception Index (ANI) method (threshold of 50/100) during phasic or tonic stimulation
  * Recording of the skin conductance reflex (skin sympathetic response) during phasic or tonic stimulations

SECONDARY OUTCOMES:
EEG time-frequency analysis during phasic pain stimulation | Day 1
  Analysis of time-frequency maps to compare the amplitude in each frequency band during phasic stimulation condition and prior baseline period
Latency of evoked responses to phasic stimulation | Day 1
  Measure of mean latency of evoked responses to phasic stimulation in a time range of 100-500 msec
Pick-to-pick amplitude of evoked responses to phasic stimulation | Day 1
  Measure of mean pick-to-pick amplitude of evoked responses to phasic stimulation in a time range of 100-500 msec
Quantification of skin sympathetic response during phasic stimulation | Day 1
  Mean area under the curve of skin sympathetic response during phasic stimulation compared to the baseline periods before stimulation
Qualitative Change of ANI Value during phasic stimulation | Day 1
  Mean percentage of decrease of ANI value during phasic stimulation compared with the baseline period before stimulation
EEG time-frequency analysis during tonic pain stimulation | Day 1
  Analysis of time-frequency maps to compare the amplitude in each frequency band during tonic stimulation condition and prior baseline period
Quantification of skin sympathetic response during tonic stimulation | Day 1
  Mean area under the curve of skin sympathetic response during tonic stimulation compared to the baseline period before stimulation
Qualitative Change of ANI Value during tonic stimulation | Day 1
  Mean percentage of decrease of ANI value during tonic stimulation compared with the baseline period before stimulation
Selection of dominant configuration of pattern in terms of sensitivity / specificity of the response to different types of nociceptive stimulation | Day 1
  Among the EEG and neurovegetative modifications, investigators will select the dominant association according to the different types of nociceptive stimulation. The dominant association will constitute the pattern of interest. This pattern will be selected if present in more than 80% of subjects. If investigators obtain several patterns of interest associating different cortical or neurovegetative parameters, the final selected pattern will be made up of the smallest number of parameters in order to envisage its transfer in anesthesiological routine

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Neurologie Fonctionnelle et Epileptologie Hôpital Neurologique, GHE Hospices civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No